CLINICAL TRIAL: NCT06300125
Title: Percutaneous Cryoablation of Low-risk Early Breast Cancer
Acronym: PRECICE
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Collaborators: Fondazione Umberto Veronesi (Other); IceCure Medical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: UID 4037; R1881/23 - L2-015 (Other: Comitato Etico Territoriale Lombardia 2)
Record Dates: First submitted 2024-02-16; First posted 2024-03-08 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Cryoablation; Ablation; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cryosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cryoablation: Percutaneous Cryoablation of Breast Cancer
  Interventions: Procedure: Cryoablation

INTERVENTIONS:
Procedure: Cryoablation — Percutaneous Cryoablation of Breast Cancer

SUMMARY:
Expand the current evidence base regarding percutaneous cryoablation of early-stage, low-risk breast tumors, integrated into the standard therapeutic pathway with well-defined follow-up data, as well as data on quality of life. Demonstrate, therefore, that the use of percutaneous cryoablation in the treatment of low-risk breast carcinoma is not inferior to surgery when combined with adjuvant radiotherapy and chemotherapy (when necessary). The hypothesis is that cryoablation, being simple and oncologically effective, ensures a better quality of life for the patient (reduced morbidity, no need for general anesthesia, improved cosmetic outcomes) and consequently has a lesser psychological impact, as well as a better cost-benefit ratio compared to the standard surgical approach.

DETAILED DESCRIPTION:
PRECICE is a prospective single arm, single centre, observational study which aims to enroll patients ≥50 years old, diagnosed with early-stage luminal A/B, unifocal Breast Cancer (BC), < 15 mm in size, without in situ component detected at imaging (by breast ultrasound, Magnetic Resonance Imaging (MRI), Mammography) and confirmed by needle biopsy, defining histotype and biology. All patients that receive treatment with cryoablation as their standard care for BC followed by RadioTherapy (RT), according to the MultiDisciplinary Tumor Board (MDTB) referral and fulfil the inclusion criteria, will be prospectively included in the study.

Follow-up protocol involved breast imaging with mammography, ultrasound, and MRI, assessment of procedure failure rate, quality of life, psychological impact, oncological outcome and economical efficacy. Adjuvant therapy will be planned after further multidisciplinary discussion

ELIGIBILITY:
Inclusion Criteria:

* Tumour, Node, Metastasis stage (TNM) = dimension up to 15 mm as measured by breast ultrasound, MRI, Mammography, Node negative, absence of distant metastasis
* Unifocality
* All invasive cancer, except lobular
* Biology= luminal A and luminal B* (Estrogen Receptor (ER) positive/human epidermal growth factor receptor-2 (HER2)negative) (Documented estrogen receptor (ER)-positive tumor assessed locally and defined as ≥10% of tumor cells stained positive.

Documented HER2-negative tumor (in accordance to 2018 American Society of Clinical Oncology guidelines, as determined per local assessment)

* Any grade (G)
* Radiological detection= breast ultrasound, MRI, Mammography
* Tumor site= not located superficially (≥1 cm from the skin plane)
* Breast size= any, appropriate for the procedure in relation to ultrasound examination
* Referral to breast cryoablation by a multidisciplinary tumor board
* Planned treatment with cryoablation using IceCure (TM-trade mark) system
* Informed consent *Luminal B and G3 BC: previous specific patients' selection and Oncotype Dx [31] on cancer tissue from needle biopsy before procedure and eventual Prediction Analysis of Microarray 50 (PAM50) test.

Exclusion Criteria:

* Plurifocality
* Invasive lobular breast cancer
* HER2 overexpressed or Triple Negative Breast Cancer (TNBC)
* tumor dimension >15 mm
* Node positive
* post NeoAdjuvant ChemoTherapy (NACT) breast cancer
* <50 years
* Presence of intraductal component (DCIS)
* Absence of psychological compliance in understanding and adhering to rationale of the study
* Inability to perform MRI
* Breast augmentation with implants

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergone percutaneous cryoablation of early stage breast cancer
Sampling Method: Probability Sample
Enrollment: 234 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Procedure failure rate | 8 months
  Percentage of patients with residual tumor at the site of cryoablation

SECONDARY OUTCOMES:
Assessment of subject's quality of life in terms of evaluation of sources of distress | 60 months
  Quality of life will be assessed using National Comprehensive Cancer Network (NCCN) DISTRESS THERMOMETER
Assessment of subject's satisfaction | 60 months
  Satisfaction will be assessed using BreastQ questionnaire
Cost-analysis - evaluation of cost of intervention, hospitalization and re-intervention (if applicable) | 60 months
  Cost will be calculated for all patients considering the cost of the intervention, the cost of hospitalization and cost of eventual re-intervention in case of unsuccessful intervention
Ipsilateral breast tumor recurrence | 60 months
  Percentage of ipsilateral breast tumor recurrence
Distant metastasis | 60 months
  Percentage of distant metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Franco Orsi, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy